CLINICAL TRIAL: NCT03205995
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of OMS721 for the Treatment of Atypical Hemolytic Uremic Syndrome (aHUS) in Adults and Adolescents
Brief Title: Safety and Efficacy Study of OMS721 in Patients With Atypical Hemolytic Uremic Syndrome
Acronym: aHUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated study
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS721-HUS-002
Expanded Access: NCT04247906 (Available)
Record Dates: First submitted 2017-04-17; First posted 2017-07-02 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome
Keywords: TMA; aHUS
MeSH Terms: conditions — Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome | interventions — narsoplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OMS721 (narsoplimab) (Experimental): Administration of OMS721 (narsoplimab)
  Interventions: Biological: OMS721 (narsoplimab)

INTERVENTIONS:
Biological: OMS721 (narsoplimab) — Intravenous loading dose followed by daily subcutaneous injections
  Other Names: narsoplimab

SUMMARY:
The purpose of this study is to evaluate the platelet count change from baseline and safety of OMS721 (narsoplimab) in adults and adolescents with atypical hemolytic uremic syndrome (aHUS). The study will also evaluate pharmacokinetics (PK), pharmacodynamics (PD), and anti-drug antibody response (ADA).

DETAILED DESCRIPTION:
This is a Phase 3, uncontrolled, open-label study to evaluate the effect of OMS721 in subjects with aHUS. The primary outcome to be measured is platelet count change from baseline. The secondary outcomes to be measured are other efficacy measures, safety, PK, PD, and immunogenicity (i.e., presence of anti-drug antibody [ADA] response. Subjects with plasma therapy-resistant aHUS and plasma therapy-responsive aHUS will be eligible. The efficacy endpoints, including the primary efficacy endpoint, may not be relevant for plasma therapy-responsive subjects because these subjects may enter the study with normal markers of aHUS activity due to successful treatment with plasma therapy. Therefore, efficacy analyses will be performed separately in the plasma therapy-resistant and plasma therapy responsive subjects. The principal efficacy analyses will be the analyses in the plasma therapy resistant cohort and efficacy analyses of the plasma therapy-responsive cohort will be supportive. Safety analyses will be conducted in all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Are age >= 12 years old at screening (Visit 1).
2. Have a primary aHUS, diagnosed clinically, and have ADAMTS13 activity > 5% in plasma. Participants are eligible with or without a documented complement mutation or anti-CFH antibody. Participants are categorized according to their response to plasma therapy (plasma exchange or plasma infusion):

   * Plasma therapy-resistant aHUS participants must have all of the following:

     * Screening platelet count < 150,000/μL despite at least four plasma therapy treatments in a 7-day period prior to screening
     * Evidence of microangiopathic hemolysis (at least one of:

       1. presence of schistocytes,
       2. serum LDH > 1.5 times upper limit of normal (ULN), and
       3. haptoglobin < LLN)
     * Serum creatinine > ULN
   * Plasma therapy-responsive aHUS participants must have all of the following:

     * Have a documented history of requiring plasma therapy to prevent aHUS exacerbation defined as all of the following:

       * decrease in platelet count > 25% when plasma therapy frequency has been decreased (including discontinuation of plasma therapy)
       * LDH > 1.5 times ULN when plasma therapy frequency has been decreased (including discontinuation of plasma therapy)
   * Have received plasma therapy at least once every 2 weeks at an unchanged frequency for at least 8 weeks before first dose of OMS721
3. If sexually active and of childbearing potential, must agree to practice a highly effective method of birth control until the end of the study, defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner.
4. Do not have access to eculizumab treatment, have not derived therapeutic benefit from eculizumab treatment, or have not been able to tolerate eculizumab treatment.

Exclusion Criteria:

1. Have STEC-HUS.
2. Have a positive direct Coombs test.
3. Have a history of hematopoietic stem cell transplant.
4. Have HUS from an identified drug.
5. History of vitamin B12 deficiency-related HUS.
6. History of Systemic Lupus Erythematosus.
7. History of antiphospholipid syndrome.
8. Active cancer or history of cancer (except non-melanoma skin cancers) within 5 years of screening.
9. Have been on hemodialysis or peritoneal dialysis for ≥ 12 weeks.
10. Have an active systemic bacterial or fungal infection requiring systemic antimicrobial therapy (prophylactic antimicrobial therapy administered as standard of care is allowed).
11. Baseline resting heart rate < 45 beats per minute or > 115 beats per minute.
12. Baseline QTcF > 470 milliseconds.
13. Have malignant hypertension (diastolic blood pressure [BP] > 120 mm Hg with bilateral hemorrhages or "cotton-wool" exudates on funduscopic examination).
14. Have a poor prognosis with a life expectancy of less than three months in the opinion of the Investigator.
15. Are pregnant or lactating.
16. Have received treatment with an investigational drug or device within four weeks of the screening visit.
17. Have abnormal liver function tests defined as ALT or AST > five times ULN.
18. Have HIV infection.
19. History of cirrhosis of the liver.
20. Are an employee of Omeros, an Investigator, a study staff member, or their immediate family member.
21. Have a known hypersensitivity to any constituent of the product.
22. Presence of any condition that the Investigator believes would put the subject at risk or confound the interpretation of the data.
23. Have previously completed treatment in an OMS721study.
24. Have received intravenous immunoglobulin (IVIG) treatment within 8 weeks of screening visit.
25. Have received rituximab within 24 weeks of screening visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Omeros Investigational Site, Chicago, Illinois, United States
- Omeros Investigational Site, Vilnius, Lithuania
- Omeros Investigational Site, Lodz, Poland
- Omeros Investigational Site, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OMS721 (Narsoplimab)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 3
  Lithuania | 3

OUTCOME MEASURES:

1. Primary Outcome: Platelet Count (10^9 Platelets/L) Change From Baseline at Week 26
Description: The primary outcome to be measured is platelet count change from baseline.
Time Frame: Week 26
Population: Any patent who received drug
Measure: Median (Full Range); unit: 10^9 platelets/L
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
10^9 platelets/L | 42 [-21 to 115.5]

2. Secondary Outcome: Safety as Measured by Incidences of Adverse Events, Vital Signs, ECG, and Clinical Laboratory Tests
Description: Assessment of safety of OMS721 (narsoplimab) in participants with aHUS by incidence of Adverse Events, clinically significant vital sign abnormalities, ECG abnormalities, and clinical laboratory test abnormalities
Time Frame: Pre-dose and up to 771 days post-dose
Population: The safety population includes all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Thrombotic Microangiopathies (TMA) Response
Description: Complete TMA response defined as normalization of platelet count, normalization of serum lactate dehydrogenase (LDH), and > 25% decrease in serum creatinine by at least 2 consecutive measures over at least 4 consecutive weeks, within the initial 26-week period
Time Frame: 26 weeks
Population: Any patient who received drug
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: TMA Event-free Status
Description: No decrease in platelet count of > 25% from baseline, no plasma exchange or plasma infusion, and no initiation of new dialysis over at least 12 consecutive weeks, within the initial 26-week period
Time Frame: 26 weeks
Population: Any patient who received drug
Measure: Count of Participants; unit: Participants
Groups:
- OMS721 (Narsoplimab): Administration of OMS721 (narsoplimab) OMS721 (narsoplimab): Intravenous loading dose followed by daily subcutaneous injections
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 2

5. Secondary Outcome: Increase in Estimated Glomerular Filtration Rate (eGFR)
Description: Increase of greater than 15 ml/min/1.73 m2 in eGFR calculated by the modification of diet in renal disease (MDRD) Equation
Time Frame: 26 weeks
Population: Any patient who received drug
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 0

6. Secondary Outcome: Hematological Normalization
Description: Normalization of platelet count and normalization of serum LDH by 2 consecutive measurements over at least 4 weeks, within the initial 26-week period
Time Frame: 26 weeks
Population: Any patient who received drug
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 1

7. Secondary Outcome: TMA Remission
Description: Platelet count greater than or equal to 150,000/μL on at least 2 consecutive measures over at least 2 consecutive weeks, within the initial 26-week period
Time Frame: 26 weeks
Population: Any patient who received drug
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 2

8. Secondary Outcome: Incidence of Antidrug Antibodies (ADA)
Description: Incidences of ADA in participants with aHUS, administered OMS721 (narsoplimab)
Time Frame: 771 days post-dose
Population: Any patient who received drug
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Participants | 1

9. Secondary Outcome: Change From Baseline in Serum Creatinine (mg/dL)
Description: Assessment of subject's change from baseline in serum creatinine.
Time Frame: 26 weeks
Population: Any patient who received drug
Measure: Median (Full Range); unit: mg/dL
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
mg/dL | 1.53 [-0.98 to 3.16]

10. Secondary Outcome: Change From Baseline in Serum LDH (U/L)
Description: Assessment of subject's change from baseline in serum LDH
Time Frame: 26 weeks
Population: Any patient who received drug.
Measure: Median (Full Range); unit: U/L
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
U/L | -12 [-112 to 389]

11. Secondary Outcome: Change From Baseline in Haptoglobin (mg/dL)
Description: Assessment of subject's change from baseline in haptoglobin
Time Frame: 26 weeks
Population: Any patient who received drug.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
mg/dL | 30 [4 to 56]

12. Secondary Outcome: Pharmacokinetics (PK): Trough Plasma Concentration, Lower Limit of Quantification (LLOQ)
Description: Pharmacokinetics (PK): Trough plasma concentration, lower limit of quantification (LLOQ)
Time Frame: Days 1-4; Treatment Maintenance (103 weeks): 17 visits; Rescue Therapy (RT) (if occurs): RT Days 1-4; Follow-Up at Day 771
Population: Pharmacokinetics trough plasma concentrations are provided on the pre-dose levels for the six patients enrolled.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
ng/mL | 15477.2 (6471.62)

13. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentrations (Cmax)
Description: Pharmacokinetics (PK): Maximum plasma concentrations (Cmax)
Time Frame: Days 1-4; Treatment Maintenance (103 weeks): 17 visits; Rescue Therapy (if occurs): RT Days 1-4; Follow-Up at Day 771
Population: The observed Cmax values on the 6 patients have been provided.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
ng/mL | 48350 [25100 to 86300]

14. Secondary Outcome: Pharmacokinetics (PK): Area Under Time-concentration Curve (AUC)
Description: Pharmacokinetics (PK): Area under time-concentration curve (AUC)
Time Frame: Days 1-4; Treatment Maintenance (103 weeks): 17 visits; Rescue Therapy (if occurs): RT Days 1-4; Follow-Up at Day 771
Population: PK modeling for calculating the AUC was not performed because the study was not completed.
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 0

15. Secondary Outcome: Pharmacodynamics (PD): Inhibition of C3 Activity (%)
Description: Pharmacodynamics (PD): Inhibition of C3 activity
Time Frame: Days 1-4; Treatment Maintenance (103 weeks): 17 visits; Rescue Therapy (if occurs): RT Days 1-4; Follow-Up at Day 771
Population: Any patient who received drug and measurable C3 activity.
Measure: Median (Full Range); unit: Inhibition of C3 activity (%)
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Inhibition of C3 activity (%) | 84.4 [1.7 to 101.4]

16. Secondary Outcome: Pharmacodynamics (PD): Inhibition of C4 Activity (%)
Description: Pharmacodynamics (PD): Inhibition of C4 activity
Time Frame: Days 1-4; Treatment Maintenance (103 weeks): 17 visits; Rescue Therapy (if occurs): RT Days 1-4; Follow-Up at Day 771
Population: Any patient who received drug and measurable C4 activity.
Measure: Median (Full Range); unit: Inhibition of C4 activity (%)
Arm/Group | OMS721 (Narsoplimab)
Number analyzed (Participants) | 6
Inhibition of C4 activity (%) | 91.9 [11.9 to 99.9]

ADVERSE EVENTS:
Time Frame: From Day 1 to Final Study Visit (up to Day 771)
Description: {Not specified}
Arm/Group | OMS721 (Narsoplimab)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMS721 (Narsoplimab) (N=6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
RENAL GRAFT INFECTION (Infections and infestations) | 2 (2)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (2)
CEREBRAL HEMATOMA (Nervous system disorders) | 1 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
HAEMOLYSIS (Blood and lymphatic system disorders) | 2 (2)
CHRONIC ALLOGRAFT NEPHROPATHY (Immune system disorders) | 1 (1)
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
ARTERIOVENOUSE FISTULA ANEURYSM (Injury, poisoning and procedural complications) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
SHUNT BLOOD FLOW EXCESSIVE (Injury, poisoning and procedural complications) | 1 (2)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (2)
Cardiac failure (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMS721 (Narsoplimab) (N=6)
BRADYCARDIA (Cardiac disorders) | 1 (2)
HAEMOLYSIS (Blood and lymphatic system disorders) | 2 (4)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (5)
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1)
INJECTION SITE EXTRAVASATION (General disorders) | 2 (2)
INJECTION SITE HAEMATOMA (General disorders) | 1 (1)
INJECTION SITE PAIN (General disorders) | 2 (3)
OEDEMA PERIPHERAL (General disorders) | 1 (2)
PYREXIA (General disorders) | 3 (4)
CHRONIC ALLOGRAFT NEPHROPATHY (Immune system disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (2)
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 1 (3)
ARTERIOVENOUS FISTULA SITE INFECTION (Infections and infestations) | 2 (2)
BACTERIAL INFECTION (Infections and infestations) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 2 (2)
MOLLUSCUM CONTAGIOSUM (Infections and infestations) | 1 (1)
RENAL GRAFT INFECTION (Infections and infestations) | 1 (1)
UREAPLASMA INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 (1)
ARTERIOVENOUS FISTULA ANEURYSUM (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
SHUNT BLOOD FLOW EXCESSIVE (Injury, poisoning and procedural complications) | 1 (2)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (4)
HUMAN CHORIONIC GONADOTROPIN ABNORMAL (Investigations) | 1 (1)
TREPONEMA TEST POSITIVE (Investigations) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (9)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 (2)
AGRESSION (Psychiatric disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (2)
HAEMATURIA (Renal and urinary disorders) | 2 (2)
LEUKOCYTURIA (Renal and urinary disorders) | 1 (1)
AMENORRHOEA (Reproductive system and breast disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (3)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (3)
Depression (Psychiatric disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT03205995/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03205995/SAP_001.pdf